CLINICAL TRIAL: NCT00556933
Title: Prospective, Randomized 2 x 2 Factorial Trial of Rabbit Anti-thymocyte Globulin Induction (Single vs. Alternate Day Administration) at Renal Transplantation, With Delayed Calcineurin-inhibitor Withdrawal vs. Minimization
Brief Title: Improved Induction and Maintenance Immunosuppression in Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0286-03-FB
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: End-stage Renal Disease
Keywords: Induction; rATG; Calcineurin-inhibitor withdrawal
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Antilymphocyte Serum; thymoglobulin; Mycophenolic Acid; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
  Interventions: Drug: rabbit anti-thymocyte globulin - single dose; Drug: sirolimus; Drug: tacrolimus
- Group 2 (Experimental): Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
  Interventions: Drug: rabbit anti-thymocyte globulin - 4 doses; Drug: sirolimus; Drug: tacrolimus
- Group 3 (Experimental): Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Interventions: Drug: rabbit anti-thymocyte globulin - single dose; Drug: mycophenolate mofetil; Drug: sirolimus; Drug: tacrolimus
- Group 4 (Experimental): Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Interventions: Drug: mycophenolate mofetil; Drug: rabbit anti-thymocyte globulin - 4 doses; Drug: sirolimus; Drug: tacrolimus

INTERVENTIONS:
Drug: rabbit anti-thymocyte globulin - single dose — A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  Other Names: Thymoglobulin; rATG
  Arms: Group 1; Group 3
Drug: mycophenolate mofetil — Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
  Other Names: CellCept; MMF; mycophenolic acid; Myfortic
  Arms: Group 3; Group 4
Drug: rabbit anti-thymocyte globulin - 4 doses — 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  Other Names: Thymoglobulin
  Arms: Group 2; Group 4
Drug: sirolimus — Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  Other Names: Rapamune, rapamycin
Drug: tacrolimus — Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
  Other Names: FK506; ProGraf

SUMMARY:
This 2 x 2 sequential factorial study evaluates two potential improvements to the standard immunosuppression regimen used at the investigators' institution to prevent rejection of transplanted kidneys. These two potential improvements are each applied in sequence to half of the study patients, creating 4 study arms; the other half receive the standard treatment. The two potential improvements are:

1. Administering the immunosuppression induction agent rATG ("rabbit anti-thymocyte globulin") in a single dose at the time of transplantation, instead of in the usual series of 4 smaller doses over 6 days.
2. After 6 months, modifying the maintenance immunosuppression used to prevent rejection by replacing the drug tacrolimus with mycophenolate mofetil (MMF).

The two interventions, spaced sequentially six months apart, enable independent analysis of the two treatments so long as it can be shown that there is no synergistic interaction between them.

DETAILED DESCRIPTION:
The two treatment innovations in this study of immunosuppression in kidney transplantation are aimed at making the transplanted kidney function sooner and last longer than is usual with standard immunosuppression regimens, but without increasing the likelihood of rejection.

The first innovation, delivering the induction agent rATG in a single large dose rather than as a series of smaller doses over 6-8 days, is expected to produce better graft function right away, possibly by reducing some of the injury to the kidney that accompanies the restoration of blood flow during transplantation ("reperfusion injury"). Some evidence has been developed by investigators elsewhere to suggest this will happen.

The second innovation, replacing tacrolimus with MMF after 6 months, is intended to eliminate a well-established major cause of ongoing toxic damage to the kidney. While tacrolimus does a good job of preventing rejection, the cost in continuing toxic injury to the kidney is high, leading inevitably to eventual graft failure, the inability of the transplanted kidney to continue filtering the blood and making adequate volumes of high-quality urine.

ELIGIBILITY:
Inclusion Criteria:

* Primary renal transplant recipient for end-stage renal disease

Exclusion Criteria:

* Recipient age < 18 years or > 65 years
* Previous history of CMV disease
* Hepatitis B and C recipients
* Primary disease states that require steroids for immunosuppression
* Re-transplant with immunological cause of renal or pancreas loss
* Non heart beating donors
* Recipient of pediatric en bloc kidneys
* Recipient with a Panel Reactive Antibody (PRA) score >75%
* Patients who have received 3 or more prior transplants, excluding pancreas
* Patients who are past recipients of other solid organ transplants
* Previous history of BK virus
* Previous treatment with Thymoglobulin
* Allergy to rabbits
* Simultaneous Kidney/Pancreas transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2011-04-01 (Actual); Study Completion 2011-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Brian Stevens, MD, PhD, Study Director — Wright State University Boonshoft School of Medicine, Dayton, OH
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Miles CD, Skorupa JY, Sandoz JP, Rigley TH, Nielsen KJ, Stevens RB. Albuminuria after renal transplantation: maintenance with sirolimus/low-dose tacrolimus vs. mycophenolate mofetil/high-dose tacrolimus. Clin Transplant. 2011 Nov-Dec;25(6):898-904. doi: 10.1111/j.1399-0012.2010.01353.x. Epub 2010 Nov 16. PMID 21077952
- [Background] Stevens RB. Modern approaches to combining sirolimus with calcineurin inhibitors. Transplant Proc. 2008 Dec;40(10 Suppl):S21-4. doi: 10.1016/j.transproceed.2008.10.012. PMID 19100901
- [Background] Sulanc E, Lane JT, Puumala SE, Groggel GC, Wrenshall LE, Stevens RB. New-onset diabetes after kidney transplantation: an application of 2003 International Guidelines. Transplantation. 2005 Oct 15;80(7):945-52. doi: 10.1097/01.tp.0000176482.63122.03. PMID 16249743
- [Result] Stevens RB, Foster KW, Miles CD, Lane JT, Kalil AC, Florescu DF, Sandoz JP, Rigley TH, Nielsen KJ, Skorupa JY, Kellogg AM, Malik T, Wrenshall LE. A randomized 2x2 factorial trial, part 1: single-dose rabbit antithymocyte globulin induction may improve renal transplantation outcomes. Transplantation. 2015 Jan;99(1):197-209. doi: 10.1097/TP.0000000000000250. PMID 25083614
- [Result] Stevens RB, Lane JT, Boerner BP, Miles CD, Rigley TH, Sandoz JP, Nielsen KJ, Skorupa JY, Skorupa AJ, Kaplan B, Wrenshall LE. Single-dose rATG induction at renal transplantation: superior renal function and glucoregulation with less hypomagnesemia. Clin Transplant. 2012 Jan-Feb;26(1):123-32. doi: 10.1111/j.1399-0012.2011.01425.x. Epub 2011 Mar 14. PMID 21401720
- [Result] Snow MH, Cannella AC, Stevens RB, Mikuls TR. Presumptive serum sickness as a complication of rabbit-derived antithymocyte globulin immunosuppression. Arthritis Rheum. 2009 Sep 15;61(9):1271-4. doi: 10.1002/art.24788. No abstract available. PMID 19714613
- [Result] Stevens RB, Mercer DF, Grant WJ, Freifeld AG, Lane JT, Groggel GC, Rigley TH, Nielsen KJ, Henning ME, Skorupa JY, Skorupa AJ, Christensen KA, Sandoz JP, Kellogg AM, Langnas AN, Wrenshall LE. Randomized trial of single-dose versus divided-dose rabbit anti-thymocyte globulin induction in renal transplantation: an interim report. Transplantation. 2008 May 27;85(10):1391-9. doi: 10.1097/TP.0b013e3181722fad. PMID 18497677
- [Derived] Stevens RB, Foster KW, Miles CD, Kalil AC, Florescu DF, Sandoz JP, Rigley TH, Malik T, Wrenshall LE. A Randomized 2x2 Factorial Clinical Trial of Renal Transplantation: Steroid-Free Maintenance Immunosuppression with Calcineurin Inhibitor Withdrawal after Six Months Associates with Improved Renal Function and Reduced Chronic Histopathology. PLoS One. 2015 Oct 14;10(10):e0139247. doi: 10.1371/journal.pone.0139247. eCollection 2015. PMID 26465152

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) (6 mg/kg) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
- Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus: Kidney transplant recipients given 4 small doses (1.5 mg/kg) of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
- Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG, 6 mg/kg x 1) and maintained on tacrolimus and sirolimus for chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
- Divided-dose rATG (1.5mg/kgx4),Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG, 1.5 mg/kg x 4) and maintained on tacrolimus and sirolimus for chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
Period: Single vs. Divided-dose rATG Induction
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG (1.5mg/kgx4),Sirolimus/Mycophenolate Mofetil
Started | 45 | 45 | 45 | 45
Completed | 43 | 37 | 39 | 43
Not Completed | 2 | 8 | 6 | 2
Not completed — Protocol Violation | 2 | 3 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Pancreas transplantation | 0 | 2 | 2 | 2
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Kidney graft primary non-function | 0 | 1 | 0 | 0
Period: CNI Withdrawal vs. Minimization
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG (1.5mg/kgx4),Sirolimus/Mycophenolate Mofetil
Started | 43 | 37 | 39 | 43
Completed | 42 | 33 | 36 | 41
Not Completed | 1 | 4 | 3 | 2
Not completed — Pancreas transplantation | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Graft loss | 0 | 1 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two patients were enrolled into the study erroneously in a violation of protocol and were identified and excluded before any study-related interventions. (Additional patients excluded from outcome analyses are accounted for in the Participant Flow and Outcome modules.)
Groups:
- Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus: Kidney transplant patients receive 6 mg/kg of rATG as a single dose administered intravenously over <24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation. Chronic maintenance immunosuppression is with tacrolimus and sirolimus.
  Sirolimus, oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  Tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
- Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus: Kidney transplant patients receive 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6. Chronic maintenance immunosuppression is with tacrolimus and sirolimus.
  Sirolimus, oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  Tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
- Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil: Kidney transplant receive the same treatment as in Group 1, until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
  Sirolimus, oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  Tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
- Divided-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofeti: Kidney transplant receive the same treatment as in Group 2, until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
  Sirolimus, oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  Tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection..
- Total: Total of all reporting groups
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofeti | Total
Number analyzed (Participants) | 44 | 44 | 45 | 45 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (12) | 47.1 (11.2) | 44.1 (13.2) | 51.6 (9.7) | 47.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 11 | 17 | 57
  Male | 29 | 30 | 34 | 28 | 121
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/Asian | 39 | 38 | 39 | 41 | 157
  Non Caucasian/Asian | 5 | 6 | 6 | 4 | 21
Patient Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (5.0) | 27.9 (6.6) | 28.8 (7.0) | 28.9 (6.9) | 28.5 (5.7)
Donor type [Number; unit: participants]
  Deceased donor | 18 | 17 | 18 | 17 | 70
  Living donor | 26 | 27 | 27 | 28 | 108
Deceased-donor Cold Ischemia Time [Mean (Standard Deviation); unit: Hours] | 14.3 (7) | 13.7 (4.1) | 14.7 (5.7) | 15.4 (11) | 14.5 (7.2)
Patient Panel Reactive Antibody (PRA)(%) [Mean (Standard Deviation); unit: % reactive] | 0.6 (2.3) | 1.0 (4.8) | 1.1 (6.3) | 1.3 (7.8) | 1.0 (5.6)
Donor/recipient height ratio [Mean (Standard Deviation); unit: ratio] | 0.98 (0.07) | 1.00 (0.17) | 0.98 (0.16) | 1.00 (0.16) | 0.99 (0.1)
Donor age [Mean (Standard Deviation); unit: years] | 40.4 (13.1) | 44.7 (10.0) | 37.4 (12.1) | 41.2 (14.0) | 40.9 (12.7)
Donor gender [Number; unit: participants]
  Male | 18 | 23 | 17 | 20 | 78
  Female | 26 | 21 | 28 | 25 | 100
Donor BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (5.7) | 27.3 (4.0) | 27.1 (4.2) | 28.3 (5.1) | 27.6 (4.8)
Donor final serum creatinine [Mean (Standard Deviation); unit: mg/dl] | 1.0 (0.3) | 1.1 (0.6) | 1.0 (0.5) | 1.0 (0.5) | 1.0 (0.5)
Adult Cadaver Donor Nyberg Grade [Mean (Standard Deviation); unit: units on a scale] — Nyberg et al (AmJourTrans 2001; 1: 162-170) developed a deceased-donor kidney grading system to predict early graft dysfunction and failure; developed from seven donor variables (cause of death, 0-6 points; history of hypertension, 0-6; final creatinine clearance before procurement, 0-6; age, 0-6; history of diabetes mellitus, 0-3; cold ischemia time, 0-3; and severity of renal artery plaque, 0-3). It stratifies deceased-donor kidneys by score: grade A, 0-5 points; grade B, 6- 10; grade C, 11-15; and grade D, 16-32. Risk of delayed graft function was 17% in Group A and 62% in group D.
  units on a scale | 10.5 (7.5) | 14.6 (7.0) | 11.8 (6.9) | 15.4 (7.8) | 13.1 (7.4)
Pediatric vs. Adult Donor [Number; unit: participants]
  Pediatric donor | 3 | 1 | 3 | 3 | 10
  Adult donor | 41 | 43 | 42 | 42 | 168
Donor/Recipient High-Risk CMV Serostatus [Number; unit: participants] — Donor/Recipient High-Risk CMV Serostatus = Donor CMV Positive/Recipient CMV Positive or Negative
  Donor/Recipient Low-Risk CMV Serostatus = Donor CMV Negative/Recipient CMV Positive or Negative
  participants
    CMV High-risk | 23 | 27 | 25 | 33 | 108
    CMV Low-risk | 21 | 17 | 20 | 12 | 70

OUTCOME MEASURES:

1. Primary Outcome: Chronic Allograft Nephropathy (Cumulative Calcineurin-inhibitor Nephrotoxicity/Transplant Nephropathy) Per Protocol Surveillance Kidney Biopsies (Banff Grading Criteria).
Description: Protocol kidney biopsies collected at approximately 12 and 24 months were scored by a transplant renal pathologist blinded to treatment group assignment for evidence of rejection, BK virus nephropathy, antibody-mediated rejection, recurrent disease, inflammation, and Banff 2005 categories of chronic renal injury. Chronic injury categories were arteriolar hyaline thickening (ah), allograft glomerulopathy (cg), interstitial fibrosis (ci), tubular atrophy (ct), and vascular fibrous intimal thickening (cv). Severity scores within each category could be 0 (<5%; none or minimal), 1 (>5% - <25%; mild), 2 (>25% - <50%, moderate), or 3 (>50%, severe). The proportions of patients in each severity grade (0, 1, 2, and 3) for both the individual categories and a composite were compared using Fisher's exact test.
Time Frame: Two years
Measure: Number; unit: percentage of participants
Groups:
- Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
  rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  sirolimus: Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
- Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
  rabbit anti-thymocyte globulin: 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  sirolimus: Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
- Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  Mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels.
- Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Rabbit anti-thymocyte globulin: 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  Mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 36 | 29 | 28 | 29
percentage of participants
  Banff histopathology cumulative grade = 0 | 43 | 40 | 53 | 51
  Banff histopathology cumulative grade = 1 | 37 | 46 | 45 | 41
  Banff histopathology cumulative grade = 2 | 16 | 9 | 2 | 7
  Banff histopathology cumulative grade = 3 | 4 | 6 | 0 | 1
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.0004, Chi-squared

2. Primary Outcome: Average of Renal Function
Description: Calculated Glomerular Filtration Rate (GFR) by using the abbreviated MDRD (aMDRD) formula and patient serum creatinine and demographic data; averaged values from months four through 24.
Time Frame: Two years
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Groups:
- Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression; tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and i
- Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression; tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
  rabbit anti-thymocyte globulin: 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  sirolimus: Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough leve
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 43 | 38 | 42 | 44
ml/min/1.73m2
  Average GFR, months 1-3 | 50.4 (16.0) | 50.1 (12.5) | 53.6 (14.4) | 50.4 (17.0)
  Average GFR, months 4-6 | 57.3 (17.6) | 57.3 (12.5) | 60.2 (15.6) | 54.8 (13.2)
  Average GFR, months 7-9 | 54.8 (16.5) | 55.0 (11.8) | 61.0 (15.8) | 55.8 (13.2)
  Average GFR, months 10-12 | 55.8 (16.6) | 55.6 (12.1) | 57.4 (16.7) | 56.6 (14.4)
  Average GFR, months 13-15 | 56.8 (19.2) | 57.3 (14.3) | 61.8 (15.4) | 58.5 (16.6)
  Average GFR, months 16-18 | 57.6 (20.9) | 56.3 (14.8) | 62.3 (17.6) | 56.6 (18.4)
  Average GFR, months 19-21 | 56.6 (20.0) | 54.8 (17.3) | 60.2 (14.7) | 56.8 (18.9)
  Average GFR, months 22-24 | 56.9 (21.9) | 57.0 (16.2) | 62.9 (18.6) | 57.6 (17.7)
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.45, General Linear Model

3. Secondary Outcome: Safety Profile
Description: Number of events: cytomegalovirus (CMV) disease, opportunistic infections (bacteremia, abscess, pneumonia, fungal), Post-transplantation Lymphoproliferative Disorder (PTLD), wound healing problems within 30 days, and lymphoceles.
Time Frame: Two years
Measure: Number; unit: Events
Units Other Than Participants: Number of possible events
Groups:
- Ingle-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  Mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels.
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Ingle-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 43 | 43 | 43 | 44
Number analyzed (Number of possible events) | 215 | 215 | 215 | 220
Events | 11 | 14 | 10 | 17
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Ingle-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.53, Fisher Exact

4. Secondary Outcome: Requirement for Additional Immunosuppression (Such as Corticosteroids, Antimetabolites or Other Immunosuppressive Agents)
Time Frame: Two years
Measure: Number; unit: participants
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 43 | 42 | 41 | 45
participants | 7 | 5 | 6 | 11
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(6mg/kg ) and Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.463, Fisher Exact

5. Secondary Outcome: Acute Rejection Per Kidney Biopsy (Banff Grading Criteria)
Time Frame: Two years
Measure: Number; unit: participants
Groups:
- Divided-dose rATG(1.5mg/kgx4), Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Rabbit anti-thymocyte globulin: 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  Mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(1.5mg/kgx4), Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 43 | 42 | 41 | 45
participants | 7 | 4 | 8 | 9
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(1.5mg/kgx4), Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.67, Kaplan-Meier

6. Secondary Outcome: Acute Tubular Necrosis (ATN) Rate, Defined as the Requirement for Dialysis Within 7 Days Post-transplantation.
Time Frame: Seven days
Measure: Number; unit: participants
Groups:
- Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Rabbit anti-thymocyte globulin: 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  Mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
Arm/Group | Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 41 | 43 | 43 | 44
participants | 3 | 1 | 6 | 2
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg x 1) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg ) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.193, Fisher Exact

7. Secondary Outcome: Graft Survival
Description: Graft failure = permanent return of patient to dialysis.
Time Frame: Two years
Measure: Number; unit: participants
Groups:
- Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
  rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  sirolimus: Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
- Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus chronic immunosuppression until tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  Rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  Mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels.
Arm/Group | Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 41 | 43 | 43 | 44
participants | 0 | 1 | 2 | 0
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.422, Fisher Exact

8. Secondary Outcome: Patient Survival
Time Frame: Two years
Measure: Number; unit: participants
Arm/Group | Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 44 | 44 | 45 | 45
participants | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.871, Fisher Exact

9. Secondary Outcome: Lymphoid Cell Sub-type CD3 Absolute Numbers
Time Frame: One year
Measure: Mean (Standard Deviation); unit: CD3 Cell Numbers/mm^3
Groups:
- Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression; tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and i
- Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression; tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
  rabbit anti-thymocyte globulin: 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  sirolimus: Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough leve
Arm/Group | Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 25 | 26 | 24 | 30
CD3 Cell Numbers/mm^3 | 446 (403) | 375 (564) | 392 (319) | 266 (211)
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.068, Kruskal-Wallis

10. Secondary Outcome: New-onset Polyomavirus (BK Virus) Disease Per Kidney Biopsy
Time Frame: Two years
Measure: Number; unit: participants
Arm/Group | Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 43 | 43 | 43 | 44
participants | 1 | 2 | 0 | 2
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.67, Fisher Exact

11. Secondary Outcome: New-onset Diabetes and Hyperglycemia After Transplantation (NODAT)
Time Frame: Six months
Measure: Number; unit: participants
Arm/Group | Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 26 | 26 | 22 | 24
participants | 10 | 7 | 5 | 12
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.21, Fisher Exact

12. Secondary Outcome: Ratio of CD4/CD8 Lymphoid Cells
Time Frame: One year
Measure: Mean (Standard Deviation); unit: Ratio of cell counts
Arm/Group | Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus | Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus | Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil | Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil
Number analyzed (Participants) | 25 | 23 | 23 | 29
Ratio of cell counts | 0.84 (0.55) | 0.84 (0.41) | 0.98 (0.53) | 1.01 (0.57)
Statistical Analysis 1: Comparison: Single Dose rATG (6 mg/kg) and Tacrolimus/Sirolimus vs Divided-dose rATG (1.5mg/kg x 4) and Tacrolimus/Sirolimus vs Single-dose rATG (6mg/kg) and Sirolimus/Mycophenolate Mofetil vs Divided-dose rATG(1.5mg/kgx4); Sirolimus/Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.40, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Up to two years.
Groups:
- Group 1: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
  rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  sirolimus: Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
- Group 2: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression.
  rabbit anti-thymocyte globulin: 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  sirolimus: Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough levels, continued indefinitely to prevent kidney rejection
  tacrolimus: Oral maintenance immunosuppressant, taken daily, dose adjusted to maintain target blood trough levels, required indefinitely to prevent kidney rejection.
- Group 3: Kidney transplant recipients given a single large dose of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression; tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  rabbit anti-thymocyte globulin: A single 6 mg/kg dose of rATG administered intravenously over 24 hours, beginning before kidney transplantation. Administration of the drug is begun as early as practical, usually after general anesthesia has been established but before surgery has started. The rATG is therefore administered for about two hours before blood flow is restored to the kidney undergoing transplantation.
  mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and i
- Group 4: Kidney transplant recipients given 4 small doses of rabbit anti-thymocyte globulin (rATG) and maintained on tacrolimus and sirolimus for chronic immunosuppression; tacrolimus is replaced with mycophenolate mofetil after about 6 months.
  mycophenolate mofetil: Patients are switched approximately 6 months after kidney transplantation from maintenance immunosuppression with tacrolimus and sirolimus to maintenance with mycophenolate mofetil and sirolimus. The drug is administered orally, taken daily, with dose adjusted in proportion to measured blood levels, and is required indefinitely to prevent rejection of the transplanted kidney.
  rabbit anti-thymocyte globulin: 6 mg/kg rabbit anti-thymocyte globulin delivered in 4 doses of 1.5 mg/kg each, the first administered at the time of kidney transplantation. Subsequent doses are administered on days 2, 4, and 6.
  sirolimus: Oral maintenance immunosuppressant administered daily, dose adjusted according to measured serum trough leve
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 9/44 | 15/44 | 18/45 | 21/45
Other Adverse Events (participants affected / at risk) | 12/44 | 12/44 | 11/45 | 8/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=44) | Group 2 (N=44) | Group 3 (N=45) | Group 4 (N=45)
Wound Abscess (Infections and infestations) | 0 | 0 | 3 | 0 — Abscess at site of transplantation incision
Wound Dehiscence (Surgical and medical procedures) | 1 | 1 | 0 | 0
Acute Tubular Necrosis (Renal and urinary disorders) | 3 | 1 | 6 | 2
Rabbit Anti-Thymocyte Globulin (rATG) Reaction (Injury, poisoning and procedural complications) | 1 | 2 | 4 | 2
Renal Allograft Primary Non-function (Renal and urinary disorders) | 0 | 1 | 0 | 0 — No or insufficient graft function from time of transplantation.
Renal Allograft Failure (Renal and urinary disorders) | 0 | 1 | 2 | 0 — Insufficient graft function necessitating permanent return to dialysis.
Ureteral Stricture (Renal and urinary disorders) | 2 | 3 | 1 | 1 — Obstruction develops in outflow tract of transplanted kidney.
Lymphocele Requiring Drainage (Surgical and medical procedures) | 3 | 1 | 2 | 4 — Failure of spontaneous resolution of lymph accumulation at site of transplanted kidney.
Repair of Wound Hernia at Transplantation Incision (Surgical and medical procedures) | 2 | 4 | 1 | 9
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1 | 1 — Myocardial infarction within 30 days of transplantation.
Cardiac Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 2 — Cardiac arrhythmia within 30 days of transplantation.
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 1
Serum Sickness (Immune system disorders) | 0 | 1 | 0 | 2 — Response to rabbit anti-thymocyte globulin administration
Death (General disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=44) | Group 2 (N=44) | Group 3 (N=45) | Group 4 (N=45)
New-onset Hyperlipidemia after Transplantation (Metabolism and nutrition disorders) | 11 | 10 | 7 | 8
Incomplete Rabbit Anti-Thymocyte Globulin Induction (Blood and lymphatic system disorders) | 1 | 2 | 4 | 0 — Administration of rabbit anti-thymocyte globulin interrupted by adverse reaction.

LIMITATIONS AND CAVEATS:
The trial is designed for analysis as 1st, rATG dosing, and 2nd, CNI withdrawal status. Results published as analysis of 2 induction protocols followed by analysis of 2 CNI maintenance regimens. Potential limitations = single-center & non-blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No